CLINICAL TRIAL: NCT04177121
Title: Qualitative Analysis Based on Medical Records of 300 Patients With Back Musculoskeletal Disorders Receiving a Physiotherapy Prescription From Primary Physicians in France
Brief Title: Qualitative Analysis of Physiotherapy Prescriptions From Primary Physicians for Patients With Back Musculoskeletal Disorders
Acronym: PresKi
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2019 / 441 CERDB
Record Dates: First submitted 2019-11-04; First posted 2019-11-26 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2020-01

CONDITIONS: Back Musculoskeletal Disorders
Keywords: Musculoskeletal disorders; Physician; Physiotherapy; Referral
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: qualitative analysis — Qualitative analysis of physiotherapy prescriptions

SUMMARY:
"Prescription in France is a major act of medical activity and must be in accordance with the scientific evidence. The use of physiotherapy by primary physicians is becoming more and more frequent and involves the performance of a prescription given to the patients so that they can access to their care. The optimization of the use of this treatment is based on the respect of several legal and regulatory provisions allowing physiotherapists (PT) to offer the most appropriate treatment to the patient. Although these professionals can carry out a physiotherapy diagnosis and the objectives of care, as well as the choice of the acts and the techniques which seem to them the most appropriate. The performance of their treatment remains conditioned by the indication to physiotherapy and the anatomical region formulated by the prescription of the primary physicians. Primary physicians don't have the right to include their diagnostic hypothesis on the physiotherapy prescription. Therefore, they could transmit to the PT a supplementary report including all useful information for the PT which could influence the progress of the treatment.

It has been reported a frequent absence of diagnostic hypothesis formulated by the primary physicians to the PT to justify the indication to these treatment with the prescription. However, PT are led to formulate one or more diagnostic hypothesis following their clinical assessment. This can lead to questioning the interest of prescription for referring the patient from the primary physician to the PT.

The qualitative study by Panchout et al shows that 97.8% of the french private physiotherapists included treat patients with musculoskeletal disorders and 95.5% received those with back disorders. Back musculoskeletal disorders are the most common conditions reported from french private PT.

No French study has yet analyzed the quality of prescriptions formulated by primary physicians for private physiotherapists. Much foreign health systems have a different model of access to physiotherapy services compared to the French system, involving direct access physiotherapy for patients with musculoskeletal disorders. This care pathway gives patients the ability to refer themselves directly to a PT without having to see another health professional. Patients do not need a prescription in this model of access to physiotherapy care to use it.

Thus, in order to optimize the relevance of the use of physiotherapy for patients with back musculoskeletal disorders, we propose a prospective and cross-sectional observational study of 60 physiotherapists. The first aim of this study is to assess the relevance of the physiotherapy indication from primary care physicians for patients with back musculoskeletal disorders and consulting physiotherapists.

DETAILED DESCRIPTION:
The main objective is to describe the contents of the documents transmitted by the primary physician to the physiotherapists relating to the physiotherapy management of patients with back musculoskeletal disorders, as well as their conformity with the results of the initial assessment of the physiotherapist.

The secondary objective is to evaluate the influence of the sociodemographic characteristics concerning the presence or the absence of diagnostic hypothesis on the primary physician documents transmitted to the physiotherapist.

The research is broken down into 9 steps:

1. Physiotherapists practicing in France will be randomly selected from the list of registered members of the National Regulatory Authority of Physiotherapists and drawn by region to obtain a representative selection of territories of these professionals,
2. The sending of patients medical records indicated to the physiotherapy for the management of a musculoskeletal condition whose prescription has been carried out by a primary physician will start from the first contacted physiotherapist who has agreed to participate in the study,
3. Each of the 60 physiotherapists contacted and who have agreed to participate in the study will meet face-to-face about the progress of the project and the anonymization of the files,
4. Physiotherapists will be asked to provide 5 medical records of patients each. The file may include: the prescription of physiotherapy given to the patient by the primary physician and / or any associated medical report transmitted to the physiotherapist by the primary physician before the start of treatment,
5. To avoid selection bias, physiotherapists will collect patient data, not opposing their participation in the study, presenting themselves consecutively with a first prescription of physiotherapy,
6. Each physiotherapist will have to anonymise on the documents: first and last name and contact information of the prescribing physician as well as the first name and the last name of the patient appearing on the prescription and associated reports. Each physiotherapist will be assigned a number (1, 2, 3, etc ...), similarly for primary physicians who prescribed physiotherapy to patients the consultant and the patients seen in consultation.

The statistical analysis will be carried out at the end of the study using SAS v9.3® Software under the responsibility of the clinical research unit.

Qualitative data will be expressed as numbers (percentage). Percentage comparisons with a Chi2 test (prescriptions without diagnostic hypothesis compared to prescriptions with diagnostic hypothesis) on the factors studied as being able to influence this criteria will be made. Comparisons of means with a non-parametric Kruskal-Wallis (or Wilcoxon) test will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18,
* Referred to a physiotherapist by a primary physician,
* Who have a prescription for physiotherapy,
* With back musculoskeletal disorders,
* Must be able to understand and speak French and legally consent to their participation in this study,
* Who did not oppose to participate in the study

Exclusion Criteria:

* Consulting the physiotherapist with a prescription for an indication other than a musculoskeletal condition of the spine
* Already taken in charge by a physiotherapist for another condition

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with back musculoskeletal disorders
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
ratio of physiotherapy prescription | 8 months
  * Indication of physiotherapy (tltled present or absent),
  * Therapeutic goals (titled present or absent),
  * Number of sessions to be performed (titled present or absent and number),
  * Anatomic region(s) to be treated (titled present or absent and region defined),
  * Physiotherapy techniques to use (titled present or absent),
  * Contraindications to physiotherapy (titled present or absent),
ratio of associated medical report | 8 months
  * Diagnostic hypothesis (present or absent),
  * Possible contraindications of certain physiotherapy techniques (present or absent).
ratio of conclusions of the physiotherapy diagnostic report | 8 months
  * Indication to physiotherapy (yes/no),
  * Diagnostic hypothesis of physiotherapists (in accordance or not with that of the prescription),
  * Compliance with the prescription concerning the number and rhythm of the sessions to be performed, the anatomical region(s) to be treated and the physiotherapy techniques to be used (in accordance or not with that of the prescription)"

SECONDARY OUTCOMES:
Self-reported assessment for sociodemographic and clinical parameters from patients with back musculoskeletal disorders and physiotherapists included | 8 months
  The assessment will be self-reported related to the sociodemographic and clinical parameters of patients with back musculoskeletal disorders influencing the quality of the prescription with the following outcomes:
  * Age,
  * Gender,
  * Residential city,
  * Pathology,
  And related to the sociodemographic and clinical parameters of physiotherapists included influencing the results of the physiotherapy diagnostic assessment:
  * Age,
  * Gender,
  * City of exercise,
  * Number of experience years,
  * Continuing education program followed in the musculoskeletal field

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie BOURMAUD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

REFERENCES:
- [Result] Demont A, Benaissa L, Recoque V, Desmeules F, Bourmaud A. Spinal pain patients seeking care in primary care and referred to physiotherapy: A cross-sectional study on patients characteristics, referral information and physiotherapy care offered by general practitioners and physiotherapists in France. PLoS One. 2022 Sep 6;17(9):e0274021. doi: 10.1371/journal.pone.0274021. eCollection 2022. PMID 36067139